CLINICAL TRIAL: NCT06501664
Title: Liposomal Irinotecan and 5-FU Versus Irinotecan / Irinotecan+5-fluorouracil as Second-line Therapy for Patients With Esophageal Squamous Cell Carcinoma: A Open-label, Randomized Study
Brief Title: Liposomal Irinotecan and 5-FU as Second-line Therapy for Patients With ESCC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rui-hua Xu, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Rui-hua Xu, MD, PhD, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-ESCC-K01
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Cancer
Keywords: liposomal irinotecan; second-line therapy; esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): liposomal irinotecan+5-FU/LV q2w
  Interventions: Drug: liposomal irinotecan; Drug: 5-FU; Drug: LV
- Control group (Active Comparator): Irinotecan q2w or irinotecan+5-FU/LV q2w
  Interventions: Drug: 5-FU; Drug: LV; Drug: Irinotecan

INTERVENTIONS:
Drug: liposomal irinotecan — Liposomal irinotecan 70 mg/m²
  Other Names: Nal-IRI
  Arms: Experimental Group
Drug: 5-FU — 5-FU 400 mg/m² bolus then 2400 mg/m2 over 46 h
  Other Names: Fluorouracil
Drug: LV — LV 400 mg/m²
  Other Names: Calcium folinate
Drug: Irinotecan — Irinotecan 180 mg/m²
  Other Names: IRI
  Arms: Control group

SUMMARY:
The aim of this study is to compare the efficacy and safety of liposome irinotecan +5-FU and irinotecan / irinotecan +5-FU regimens in the second-line treatment of esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
Esophageal cancer was ranked the sixth most common cancer worldwide and seventh most common cause of cancer-related deaths. ESCC is the most common histologic subtype in Asia. The National Comprehensive Cancer Network (NCCN) guidelines recommend immune checkpoint inhibitors, taxanes, fluorouracils and/or irinotecan as the second-line treatment of ESCC. Liposomal irinotecan is a new pharmaceutical form of traditional irinotecan. It adopts a special loading technology to encapsulate traditional irinotecan in liposomes, which can avoid its hydrolysis under physiological conditions, increase the affinity with cancer cells, overcome drug resistance, increase the drug uptake by cancer cells, reduce the drug dose, improve the efficacy and reduce the toxic side effects. The aim of this study is to compare the efficacy and safety of liposome irinotecan +5-FU and irinotecan / irinotecan +5-FU regimens in the second-line treatment of esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old.
* Unresectable esophageal squamous cell carcinoma confirmed by histopathology and/or cytology.
* Failure or intolerance to first-line treatment.
* At least one measurable lesion (according to RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1.
* The expected survival time ≥3 months.
* Subject has adequate biological parameters as demonstrated by the following: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin (Hgb) ≥90 g/L.
* Adequate hepatic function as evidenced by total bilirubin ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN, ≤5 x ULN if liver metastases are present. Documented serum albumin ≥ 3 g/dL.
* Adequate renal function as evidenced by serum creatinine (Cr)≤1.5 x ULN or creatinine clearance ≥60 mL/min.
* Subjects agree to use contraception and are not pregnant or breastfeeding women.
* Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening.

Exclusion Criteria:

* Any other malignancy within 5 years prior to randomization, with the exception of cured in-situ carcinoma or basal cell carcinoma.
* Received irinotecan/irinotecan liposome based therapy in the first line.
* Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
* Active HIV infection.
* Combined with uncontrollable systemic diseases, such as unstable angina, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmia, severe pericardial disease history and other cardiovascular diseases; uncontrolled hypertension(Defined as systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90 mmHg after treatment with standardized antihypertensive drugs), or history of critical hypertension, hypertensive encephalopathy; uncontrollable diabetes, etc.
* Presence of severe gastrointestinal disease (including active bleeding, > grade 1 obstruction , > grade 1 diarrhea or gastrointestinal perforation)
* Allergy to or intolerance to therapeutic drugs or their excipients.
* Presence of central nervous system metastasis.
* Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1.
* Participated in other trial within 30 days or within 5 half-lives of the drug prior to the first dose of study treatment.
* Patients who are not suitable to participate in this trial for any reason judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Defined as the time between the date of randomization and death due to various causes

SECONDARY OUTCOMES:
Objective Response Rate | 4 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1
Disease Control Rate | 4 months
  Defined as the percentage of patients who achieved CR, PR, and stable disease (SD) according to RECIST v1.1
Progress-free survival | 5 months
  Defined as time from the date of randomization to first documented disease progression using RECIST version 1.1 by investigator review or death due to any cause, whichever occurred first.
Incidence of adverse events | 5 months
  Use NCI-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Professor, Principal Investigator — Yat-sen University Cancer Center

IPD SHARING:
Plan to Share IPD: No